CLINICAL TRIAL: NCT06136442
Title: Atogepant in Real Life in Italy
Brief Title: Atogepant in Real Life in Italy (GIANT)
Acronym: GIANT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Other Study IDs: IRCCS San Raffaele
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-01

CONDITIONS: Migraine, Prophylaxis
MeSH Terms: conditions — Migraine Disorders | interventions — atogepant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Atogepant — atogepant in real life in Italy

SUMMARY:
Atogepant is an oral, small-molecule, calcitonin gene-related peptide (CGRP) receptor antagonist that has been approved for the preventive treatment of episodic and chronic migraine (>= 4 monthly migraine days) with or without medication overuse.

DETAILED DESCRIPTION:
This study is designed to confirm the effectiveness and safety of atogepant in real life. The primary endpoint is the change from baseline in the mean number of monthly migraine days (MMDs)across the 12 weeks. Secondary endpoints include: change in monthly analgesic intake, Numeric Rating Scale (NRS), Headache Impact Test-6 (HIT-6) and Migraine disability assessment (MIDAS) scores, >=50%, >=75%, 100% responders, >=50%, >=75%, 100% responders in patients with medication overuse at weeks 9-12 compared to baseline and adverse events eventually occur during 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria: •

Age: >18 yrs Diagnosis of migraine Migraine frequency: >=4 monthly migraine days (MMDs)

Exclusion Criteria:

Patients using concomitant migraine prophylaxis Use of onabotulinumtoxinA during the previous 12 weeks Exposure to anti-CGRP mAbs during the previous 24 weeks Clinically significant cardiovascular disorders

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: migraine patients with >=4 monthly migraine days (MMDs)
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04-09 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in monthly migraine days at weeks 9-12 compared to baseline | 12 weeks
  variation of number of monthly migraine days

SECONDARY OUTCOMES:
Change in monthly analgesic intake at weeks 9-12 compared to baseline | 12 weeks
  variation of number of analgesic intake
Change in Numerical Rating Scale (NRS) score at weeks 9-12 compared to baseline | 12 weeks
  variation of Numerical Rating Scale (NRS) score
Change in HIT-6 (Headache Impact Test) score at weeks 9-12 compared to baseline | 12 weeks
  variation of HIT-6
Change in Migraine Disability Assessment Test Score (MIDAS) at weeks 1-12 compared to baseline Change in MIDAS (Migraine Disability Assessment Score) score at weeks 9-12 compared to baseline | 12 weeks
  variation of MIDAS
>50%, >75%, 100% responders at weeks 9-12 compared to baseline | 12 weeks
  proportion of migraine patients who respond to atogepant with reduction of MMDs >=50%, >=75% and 100%
>50%, >75%, 100% responders at weeks 9-12 compared to baseline in patients with Medication overuse | 12 weeks
  proportion of migraine patients with medication overuse who respond to atogepant with reduction of MMDs >=50%, >=75% and 100%
adverse events | 12 weeks
  adverse events eventually occur during 12 weeks of treatment

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goadsby PJ, Dodick DW, Ailani J, Trugman JM, Finnegan M, Lu K, Szegedi A. Safety, tolerability, and efficacy of orally administered atogepant for the prevention of episodic migraine in adults: a double-blind, randomised phase 2b/3 trial. Lancet Neurol. 2020 Sep;19(9):727-737. doi: 10.1016/S1474-4422(20)30234-9. PMID 32822633
- [Result] Min KC, Kraft WK, Bondiskey P, Colon-Gonzalez F, Liu W, Xu J, Panebianco D, Mixson L, Dockendorf MF, Matthews CZ, Boinpally R. Atogepant Is Not Associated With Clinically Meaningful Alanine Aminotransferase Elevations in Healthy Adults. Clin Transl Sci. 2021 Mar;14(2):599-605. doi: 10.1111/cts.12917. Epub 2020 Nov 24. PMID 33142014
- [Result] Ailani J, Lipton RB, Goadsby PJ, Guo H, Miceli R, Severt L, Finnegan M, Trugman JM; ADVANCE Study Group. Atogepant for the Preventive Treatment of Migraine. N Engl J Med. 2021 Aug 19;385(8):695-706. doi: 10.1056/NEJMoa2035908. PMID 34407343